CLINICAL TRIAL: NCT04830748
Title: Effect of Mechanical Traction and Therapeutic Exercises in Treatment of Primary Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, moaaz ragab riyad amin, Teaching assistant at faculty of physical therapy, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MT & TE & 1ry KOA
Record Dates: First submitted 2021-03-19; First posted 2021-04-05 (Actual); Last update posted 2022-12-08 (Actual); Status verified 2022-12

CONDITIONS: Knee Osteoarthritis
Keywords: Traction; Distraction; Therapeutic exercises
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Exercise Therapy

STUDY DESIGN:
Intervention Model Description: 2 groups
  The first group will include 20 patients and will receive therapeutic exercises in the form of stretching and strengthening exercises of the knee.
  The second group will include 20 patients and will receive the same exercise program of the first group preceded by continuous mechanical traction of the knee.
Who Masked: Participant, Outcomes Assessor
Masking Description: Patients will be blinded to study hypotheses and informed only about comparing different programs of treatment of knee osteoarthritis. After randomization, participants will only be provided with details of the program they will be undertaking.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Therapeutic exercises group (Active Comparator): The first group will receive therapeutic exercises in the form of stretching and strengthening exercises of the knee.
  Interventions: Other: Therapeutic exercises
- Therapeutic exercises and mechanical traction group (Experimental): The experimental group will receive the same exercise program of the first group preceded by continuous mechanical traction of the knee.
  Interventions: Other: Mechanical knee traction; Other: Therapeutic exercises

INTERVENTIONS:
Other: Mechanical knee traction — Continuous knee joint mechanical traction will be applied to the patients positioned in supine lying position with the affected knee flexed at 25-30 degrees by a wedge placed under the affected knee. The thigh will be secured with a strap for stabilization and the leg will be held by the specially designed greave with the weight of traction hanging throughout a pulley system. The amount of traction will be set to about 10% of body weight. The treatment will be applied for 20 minutes continuously, once a day, 3 times per week for 4 weeks. The traction force will be progressed gradually during the program ( e.g.: weekly increase force by 1% of body weight if the patient can tolerate the duration of 20 min with the preset force).
  Arms: Therapeutic exercises and mechanical traction group
Other: Therapeutic exercises — Therapeutic exercises will be divided into stretching and strengthening exercises:
  Stretching will be done passively for the hamstring, rectus femoris and calf muscles. Each exercise will be done for 3 reps each with a hold period of 30-60 secs with a 30-60 rest period between reps.
  Strengthening exercises will be done for the quadriceps and hamstring muscles ( inner range knee extension- knee extension in sitting- straight leg raise in flexion- prone hamstring curl- standing hamstring curl- straight leg raise in extension). Exercise will be done for 3 sets each will consist of 10 reps with a rest period of 2-3 minutes between sets. The starting weight should be 50% of the patient's 1 RM. The end position will be held for 5 seconds. Progression will be achieved by increasing the exercise rep and intensity gradually throughout the program. E.g.: weekly increase force by 5% if patient can tolerate an increased repetition of 20 rep with the preset force.

SUMMARY:
The purpose of this study is to compare between therapeutic exercises and therapeutic exercises preceded by mechanical traction in treatment of patients with primary knee osteoarthritis attributed to the outcomes of pain, muscle strength, functional disability and functional performance.

Hypotheses

1. There will be no significant difference between therapeutic exercises and therapeutic exercises preceded by mechanical traction on reduction of knee pain severity in patients with primary knee osteoarthritis.
2. There will be no significant difference between therapeutic exercises and therapeutic exercises preceded by mechanical traction on reduction of functional disability in patients with primary knee osteoarthritis.
3. There will be no significant difference between therapeutic exercises and therapeutic exercises preceded by mechanical traction on increasing isometric quadriceps muscle strength in patients with primary knee osteoarthritis.
4. There will be no significant difference between therapeutic exercises and therapeutic exercises preceded by mechanical traction on increasing isometric hamstring muscle strength in patients with primary knee osteoarthritis.
5. There will be no significant difference between therapeutic exercises and therapeutic exercises preceded by mechanical traction on decreasing walking time in patients with primary knee osteoarthritis.
6. There will be no significant difference between therapeutic exercises and therapeutic exercises preceded by mechanical traction on decreasing ascending and descending stairs time in patients with primary knee osteoarthritis.

DETAILED DESCRIPTION:
Knee osteoarthritis is the most common cause of musculoskeletal pain and disability, resulting in major disability and pain in affected individuals. It is a chronic degenerative disorder of multifactorial aetiology, including acute and/or chronic insults from normal wear and tear, age, obesity and joint injury. It nearly affects about one in each eight adults worldwide, its prevalence rates vary from 7.8 to 9.3% in Egyptian population.

Current clinical guidelines recommend non pharmacological conservative strategies including physical therapy given their ease of application and relatively low cost with minimal adverse effects (e.g.: strengthening exercises, aerobic exercises, stretching exercises, hydrotherapy, manual therapy, massage therapy, thermotherapy, electrotherapy, ultrasound therapy, external support braces and taping).

It was reported that therapeutic exercise is beneficial for patients with knee osteoarthritis in terms of outcomes of pain, function, performance and quality of life. In addition, it was reported that strengthening, flexibility and neuromotor skill exercises have a large efficacy over aerobic and mind body exercise.

Unloading strategies should be proposed as a first line of therapy for the patient with knee osteoarthritis before any attempts are made at tissue regeneration, repair or replacement.

Manual or mechanical knee joint distraction is a conservative technique that provides transient joint separation and unloading that aids in improving clinical symptoms of patients.

Addition of mechanical knee distraction to therapeutic exercises helps in gaining the positive effects of both exercise and unloading techniques. Although this approach has not been used extensively or applied pragmatically, several studies were found showing promising results in terms of reducing pain at both rest and movement, improving knee flexion and extension range of motion, reducing disability, increasing functional abilities and improving the quality of life of patients.

Forty male and female patients with the diagnosis of primary knee osteoarthritis will be recruited in this study. All patients will be assessed and treated in the outpatient clinic of the faculty of physical therapy, Cairo University. Patients will be randomly distributed into 2 equal experimental groups: the first experimental group will receive therapeutic exercises (stretching and strengthening exercise) while the second experimental group will receive mechanical traction of the knee followed by therapeutic exercises. All patients will be treated for 12 sessions, 3 times per week each other day for 4 weeks. Clinical assessments will include assessment of pain severity, functional disability, isometric muscle strength, and functional performance.

ELIGIBILITY:
Inclusion Criteria:

* Patients will have grade II of primary knee osteoarthritis.
* Patients with bilateral primary knee osteoarthritis, the more painful knee will be selected as the affected knee in this study.
* Age of patients will range from 45 years to 65 years old.
* Duration of illness will range from 3- 12 months.

Exclusion Criteria:

* Malignancy
* presence of skin lesions or infections at the treatment sites

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Measurement of knee pain severity change after 4 weeks of intervention | baseline, 4 weeks
  Knee pain severity will be measured on an 11-point numerical pain rating scale, where 0= no pain and 10= worst possible pain.

SECONDARY OUTCOMES:
Measurement of Functional Disability change after 4 weeks of intervention | baseline, 4 weeks
  The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) is a self-administered patient reported measure that is both valid and disease-specific.It has been translated and validated into Arabic language. It is a 24-item questionnaire, grouped into three subscales including pain; stiffness; and physical function. Total score ranges from 0 (best) to 96 (worst) points.
Measurement of Isometric quadriceps and hamstring Muscle Strength change after 4 weeks of intervention | baseline, 4 weeks
  Isometric muscle strength (Nm/kg) will be recorded for quadriceps and hamstring muscle groups. Using a hand held dynamo-meter the torque generated by the muscle is measured in newton-metre (Nm) which is later normalised to body mass in kilograms (kg).
  muscle strength = Torque (Nm) / body mass (kg).
Measurement of Functional Performance change after 4 weeks of intervention using the 40 meter fast paced walk test | baseline, 4 weeks
  The 40 meter fast paced walk test is a performance-based test that measures short distance walking activity. Three trials will be done for each test with a 5 min. rest between trials and a 10 min. rest between tests.
Measurement of Functional Performance change after 4 weeks of intervention using the 12 step stair climb test | baseline, 4 weeks
  The 12 step stair climb test is a performance-based test that measures the time required to go up and down 12 stairs (step height, 17 cm; step depth, 30 cm). Three trials will be done for each test with a 5 min. rest between trials and a 10 min. rest between tests.

CONTACTS AND LOCATIONS:
Overall Officials: Karima Abdelaty Hassan, lecturer, Study Director — Cairo University; Ibrahim Magdy Elnaggar, Prof, Study Director — Cairo University
Locations (1):
- Faculty of physical therapy Cairo university, Cairo, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alpayci M, Ozkan Y, Yazmalar L, Hiz O, Ediz L. A randomized controlled trial on the efficacy of intermittent and continuous traction for patients with knee osteoarthritis. Clin Rehabil. 2013 Apr;27(4):347-54. doi: 10.1177/0269215512459062. Epub 2012 Sep 7. PMID 22960239
- [Background] Bellamy N, Campbell J, Stevens J, Pilch L, Stewart C, Mahmood Z. Validation study of a computerized version of the Western Ontario and McMaster Universities VA3.0 Osteoarthritis Index. J Rheumatol. 1997 Dec;24(12):2413-5. PMID 9415651
- [Background] Bohannon RW. Measuring knee extensor muscle strength. Am J Phys Med Rehabil. 2001 Jan;80(1):13-8. doi: 10.1097/00002060-200101000-00004. PMID 11138949
- [Background] Brosseau L, Taki J, Desjardins B, Thevenot O, Fransen M, Wells GA, Mizusaki Imoto A, Toupin-April K, Westby M, Alvarez Gallardo IC, Gifford W, Laferriere L, Rahman P, Loew L, De Angelis G, Cavallo S, Shallwani SM, Aburub A, Bennell KL, Van der Esch M, Simic M, McConnell S, Harmer A, Kenny GP, Paterson G, Regnaux JP, Lefevre-Colau MM, McLean L. The Ottawa panel clinical practice guidelines for the management of knee osteoarthritis. Part two: strengthening exercise programs. Clin Rehabil. 2017 May;31(5):596-611. doi: 10.1177/0269215517691084. Epub 2017 Feb 1. PMID 28183213
- [Background] Chopra A, Abdel-Nasser A. Epidemiology of rheumatic musculoskeletal disorders in the developing world. Best Pract Res Clin Rheumatol. 2008 Aug;22(4):583-604. doi: 10.1016/j.berh.2008.07.001. PMID 18783739
- [Background] Fransen M, McConnell S, Harmer AR, Van der Esch M, Simic M, Bennell KL. Exercise for osteoarthritis of the knee: a Cochrane systematic review. Br J Sports Med. 2015 Dec;49(24):1554-7. doi: 10.1136/bjsports-2015-095424. Epub 2015 Sep 24. PMID 26405113
- [Background] Guermazi A, Hunter DJ, Roemer FW. Plain radiography and magnetic resonance imaging diagnostics in osteoarthritis: validated staging and scoring. J Bone Joint Surg Am. 2009 Feb;91 Suppl 1:54-62. doi: 10.2106/JBJS.H.01385. PMID 19182026
- [Background] Guermazi M, Poiraudeau S, Yahia M, Mezganni M, Fermanian J, Habib Elleuch M, Revel M. Translation, adaptation and validation of the Western Ontario and McMaster Universities osteoarthritis index (WOMAC) for an Arab population: the Sfax modified WOMAC. Osteoarthritis Cartilage. 2004 Jun;12(6):459-68. doi: 10.1016/j.joca.2004.02.006. PMID 15135142
- [Background] Kennedy DM, Stratford PW, Wessel J, Gollish JD, Penney D. Assessing stability and change of four performance measures: a longitudinal study evaluating outcome following total hip and knee arthroplasty. BMC Musculoskelet Disord. 2005 Jan 28;6:3. doi: 10.1186/1471-2474-6-3. PMID 15679884
- [Background] Khademi-Kalantari K, Mahmoodi Aghdam S, Akbarzadeh Baghban A, Rezayi M, Rahimi A, Naimee S. Effects of non-surgical joint distraction in the treatment of severe knee osteoarthritis. J Bodyw Mov Ther. 2014 Oct;18(4):533-9. doi: 10.1016/j.jbmt.2013.12.001. Epub 2013 Dec 11. PMID 25440203
- [Background] Lee DK, Lee NY. Case study of continuous knee joint traction treatment on the pain and quality of life of patients with degenerative gonarthritis. J Phys Ther Sci. 2018 Jun;30(6):848-849. doi: 10.1589/jpts.30.852. Epub 2018 Jun 12. PMID 29950778
- [Background] Maher S, Creighton D, Kondratek M, Krauss J, Qu X. The effect of tibio-femoral traction mobilization on passive knee flexion motion impairment and pain: a case series. J Man Manip Ther. 2010 Mar;18(1):29-36. doi: 10.1179/106698110X12595770849560. PMID 21655421
- [Background] McAlindon TE, Bannuru RR, Sullivan MC, Arden NK, Berenbaum F, Bierma-Zeinstra SM, Hawker GA, Henrotin Y, Hunter DJ, Kawaguchi H, Kwoh K, Lohmander S, Rannou F, Roos EM, Underwood M. OARSI guidelines for the non-surgical management of knee osteoarthritis. Osteoarthritis Cartilage. 2014 Mar;22(3):363-88. doi: 10.1016/j.joca.2014.01.003. Epub 2014 Jan 24. PMID 24462672
- [Background] Palhais NS, Guntern D, Kagel A, Wettstein M, Mouhsine E, Theumann N. Direct magnetic resonance arthrography of the knee: utility of axial traction. Eur Radiol. 2009 Sep;19(9):2225-31. doi: 10.1007/s00330-009-1389-3. Epub 2009 Apr 7. PMID 19350249
- [Background] Rausch Osthoff AK, Niedermann K, Braun J, Adams J, Brodin N, Dagfinrud H, Duruoz T, Esbensen BA, Gunther KP, Hurkmans E, Juhl CB, Kennedy N, Kiltz U, Knittle K, Nurmohamed M, Pais S, Severijns G, Swinnen TW, Pitsillidou IA, Warburton L, Yankov Z, Vliet Vlieland TPM. 2018 EULAR recommendations for physical activity in people with inflammatory arthritis and osteoarthritis. Ann Rheum Dis. 2018 Sep;77(9):1251-1260. doi: 10.1136/annrheumdis-2018-213585. Epub 2018 Jul 11. PMID 29997112
- [Background] Sato T, Sato N, Masui K, Hirano Y. Immediate effects of manual traction on radiographically determined joint space width in the hip joint. J Manipulative Physiol Ther. 2014 Oct;37(8):580-5. doi: 10.1016/j.jmpt.2014.08.002. Epub 2014 Sep 4. PMID 25200270
- [Background] Waller C, Hayes D, Block JE, London NJ. Unload it: the key to the treatment of knee osteoarthritis. Knee Surg Sports Traumatol Arthrosc. 2011 Nov;19(11):1823-9. doi: 10.1007/s00167-011-1403-6. Epub 2011 Feb 5. PMID 21298256